CLINICAL TRIAL: NCT04524897
Title: The Use of Triamcinolone Injection in Treatment of Refractory Benign Esophageal Stricture in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Zuhry, assiut university children hospital, assistant lecturer ,gastroentrologyand hepatology and endoscopy unit., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIRBESC
Record Dates: First submitted 2020-08-16; First posted 2020-08-24 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Stricture
Keywords: triamcinolole; refractory esophageal stricture; children
MeSH Terms: conditions — Esophageal Stenosis | interventions — Triamcinolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The use of Triamcinolone Injection (Other): Triamcinolone acetate (40 mg/mL)
  Interventions: Drug: Triamcinolone Injection in treatment of refractory benign Esophageal Stricture in children

INTERVENTIONS:
Drug: Triamcinolone Injection in treatment of refractory benign Esophageal Stricture in children — Triamcinolone Injection in treatment of refractory benign Esophageal Stricture with endoscopic dilatation
  Other Names: Triamcinolone Injection in treatment of refractory benign Esophageal Stricture with endoscopic dilatation

SUMMARY:
To evaluate the efficacy of Intra-lesional triamcinolone injection in the management of refractory benign esophageal Stricture in children.

DETAILED DESCRIPTION:
Oesophageal stricture is a commonly encountered clinical problem, especially in gastroenterology. It occurs due to narrowing of oesophagus, which results in swallowing difficulty. Oesophageal stricture has two major types: benign and malignant. Malignant type results from carcinoma but benign type has different causes.

Amongst benign aetiologies, gastrointestinal reflux disease (GERD), peptic injury, oesophageal webs, radiation damage, caustic swallowing and anastomotic strictures are most common. Corrosive intake is an important public health issue in developed countries and its incidence is still increasing in developing countries. The problem is largely unreported and its exact prevalence cannot be figured out due to the insufficient reporting or personal experience.

Corrosives materials can damage the bodies' tissues, as they come in contact with them. They are usually utilised to clean metals. It can cause severe health hazard, if swallowed accidentally or intentionally. Epidemiological studies have documented corrosive intake as the third most common cause of poisoning in adults.

The most common symptom of oesophageal stricture is progressive dysphagia to solids followed by inability to tolerate liquids. These strictures are diagnosed most commonly by using barium swallow, endoscopy and biopsy. Endoscopic dilatation is the most applicable method to treat oesophageal strictures, and proton pump inhibitors (PPIs) are also used to inhibit acid production.

According to the Kochman criteria, refractory or recurrent strictures are defined as an anatomic restriction because of a cicatricial luminal compromise or fibrosis resulting in clinical symptoms of dysphagia in the absence of endoscopic evidence of inflammation. This may occur as the result of either an inability to successfully remediate the anatomic problem to a diameter of at least 14 mm over five sessions at two-week intervals (refractory); or as a result of an inability to maintain a satisfactory luminal diameter for four weeks once the target diameter of 14 mm has been achieved (recurrent). This definition is not meant to include patients with an inflammatory stricture (which will not resolve until the inflammation subsides), or those with a satisfactory diameter but having dysphagia on the basis of neuromuscular dysfunction (for example those with dysphagia due to postoperative and/or postradiation therapy).

Esophageal rehabilitation has been carried out for many years with different techniques, depending on the experience of each physician, esophageal prostheses or splints, dilations with balloons or Savary-Gilliard plugs, Hurst dilators, etc., have been used, but in reality, there is no worldwide standardization for the management of these patients and even less so for the use of certain substances such as triamcinolone acetonide applied intralesionally, or more recently, topical mitomycin C.

Triamcinolone acetonide is a synthetic corticosteroid with a preventive effect on collagen synthesis, fibrosis, and chronic cicatrization that has been used for many years, applied in intralesional injection after esophageal dilations for the purpose of delaying cicatrization and thus reducing the number of dilations.

Presently, through many studies, it has been concluded that intralesional corticosteroid injections can be added to standard treatment for corrosive oesophageal stricture. International literature exhibited that intralesional steroid injections help in increasing the diameter because of its anti-inflammatory action.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Assiut University Children Hospital with:
* refractory benign esophageal stricture(inability to successfully remediate the anatomic problem to a diameter of at least 14 mm over five sessions at two-week interval)
* inability to maintain a satisfactory luminal diameter for four weeks once the target diameter of 14 mm has been achieved

Exclusion Criteria:

* Pharyngeal stenosis precluding endoscopic examination and dilatation
* tracheo-esophageal fistula,
* gastric cicatrization that precluded safe placement of aguidewire
* any patient who was unfit for general anesthesia.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
number of patients show improvement in dysphagia scale after five session of triamcinolone injection | 2years
  number of patients show improvement in dysphagia scale after five session of triamcinolone injection

SECONDARY OUTCOMES:
the number of patients who will show complete relieve of dysphagia after five sessions of triamcinolone injection | 2years
  complete abscence of dysphagia after triamcinolone injection

CONTACTS AND LOCATIONS:
Overall Officials: Nagla Abou Faddan, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Morikawa N, Honna T, Kuroda T, Watanabe K, Tanaka H, Takayasu H, Fujino A, Tanemura H, Matsukubo M. High dose intravenous methylprednisolone resolves esophageal stricture resistant to balloon dilatation with intralesional injection of dexamethasone. Pediatr Surg Int. 2008 Oct;24(10):1161-4. doi: 10.1007/s00383-008-2224-7. PMID 18704454
- [Background] Contini S, Scarpignato C. Caustic injury of the upper gastrointestinal tract: a comprehensive review. World J Gastroenterol. 2013 Jul 7;19(25):3918-30. doi: 10.3748/wjg.v19.i25.3918. PMID 23840136
- [Background] Mowry JB, Spyker DA, Cantilena LR Jr, McMillan N, Ford M. 2013 Annual Report of the American Association of Poison Control Centers' National Poison Data System (NPDS): 31st Annual Report. Clin Toxicol (Phila). 2014 Dec;52(10):1032-283. doi: 10.3109/15563650.2014.987397. PMID 25559822
- [Background] Park KS. Evaluation and management of caustic injuries from ingestion of Acid or alkaline substances. Clin Endosc. 2014 Jul;47(4):301-7. doi: 10.5946/ce.2014.47.4.301. Epub 2014 Jul 28. PMID 25133115
- [Background] Kochman ML, McClave SA, Boyce HW. The refractory and the recurrent esophageal stricture: a definition. Gastrointest Endosc. 2005 Sep;62(3):474-5. doi: 10.1016/j.gie.2005.04.050. No abstract available. PMID 16111985
- [Background] Berger M, Ure B, Lacher M. Mitomycin C in the therapy of recurrent esophageal strictures: hype or hope? Eur J Pediatr Surg. 2012 Apr;22(2):109-16. doi: 10.1055/s-0032-1311695. Epub 2012 Apr 19. PMID 22517516
- [Background] Ravich WJ. Endoscopic Management of Benign Esophageal Strictures. Curr Gastroenterol Rep. 2017 Aug 24;19(10):50. doi: 10.1007/s11894-017-0591-8. PMID 28840483
- [Background] Nagaich N, Nijhawan S, Katiyar P, Sharma R, Rathore M. Mitomycin-C: 'a ray of hope' in refractory corrosive esophageal strictures. Dis Esophagus. 2014 Apr;27(3):203-5. doi: 10.1111/dote.12092. Epub 2013 Jun 24. PMID 23796367
- [Background] Poddar U, Thapa BR. Benign esophageal strictures in infants and children: results of Savary-Gilliard bougie dilation in 107 Indian children. Gastrointest Endosc. 2001 Oct;54(4):480-4. doi: 10.1067/mge.2001.118253. PMID 11577311